CLINICAL TRIAL: NCT06743269
Title: Time-efficient Inspiratory Muscle Strength Training for Improving Sympathetic Activity, Hot Flashes, and Sleep in Midlife Women
Brief Title: Improving Sympathetic Activity, Hot Flashes, and Sleep in Midlife Women Using Inspiratory Muscle Strength Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sarah E. Baker, Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 23-011042
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Menopause; Hot Flashes; Blood Pressure Regulation
Keywords: menopause; blood pressure; inspiratory training; hot flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Resistance Inspiratory Muscle Strength Training Group (Experimental): Subjects will partake in 5 sets of 6 inspiratory maneuvers (total: 30 maneuvers/session) 6 days a week for 6 weeks using the POWERbreathe K3 device to monitor adherence.
  Interventions: Behavioral: High-Resistance Inspiratory Muscle Strength Training; Device: POWERbreathe K3 device
- Low-Resistance Inspiratory Muscle Strength Training Group (Active Comparator): Subjects will partake in 5 sets of 6 inspiratory maneuvers (total: 30 maneuvers/session) 6 days a week for 6 weeks using the POWERbreathe K3 device to monitor adherence.
  Interventions: Behavioral: Low-Resistance Inspiratory Muscle Strength Training; Device: POWERbreathe K3 device

INTERVENTIONS:
Behavioral: High-Resistance Inspiratory Muscle Strength Training — Performs inspiratory maneuvers at 55% maximal inspiratory pressure (PIMAX) during week 1, 65% PIMAX during week 2, and 75% PIMAX during weeks 3-6.
  Arms: High-Resistance Inspiratory Muscle Strength Training Group
Behavioral: Low-Resistance Inspiratory Muscle Strength Training — Performs inspiratory maneuvers at 15% maximal inspiratory pressure (PIMAX) for all 6 weeks.
  Arms: Low-Resistance Inspiratory Muscle Strength Training Group
Device: POWERbreathe K3 device — Inspiratory muscle training device

SUMMARY:
The purpose of this research is to understand how training the muscles used for breathing (inhalation) affects menopausal hot flashes, sympathetic nerve activity and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 45-60 with hot flashes.
* Participants will be recruited from Rochester, MN and surrounding areas.
* Non-smokers.
* BMI < 40kg/m^2.
* No history of cardiovascular disease, except for hypertension.

Exclusion Criteria:

* Detailed medical and social histories will be collected. To allow for ecological validity, participants will not be excluded for use of menopausal hormone therapy or medications affecting cardiovascular function so long as they have been on a consistent regimen for ≥3 months and during the study period. This approach to medications is consistent with recent work in this area.
* Participants will be screened for contraindications to inspiratory muscle strength training including, a history of spontaneous pneumothorax, collapsed lung that has not healed fully, a perforated eardrum that has not healed fully, and/or any other condition of the eardrum.
* Additional exclusion criteria will include the use of sleep aids (i.e., prescription, melatonin, doxylamine, valerian root, etc.).

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline, 6 weeks
  Measured in millimeters of mercury (mm Hg)
Change in Muscle Sympathetic Nerve Activity (MSNA) burst frequency | Baseline, 6 weeks
  Measured by microneurography reported in burst per minute
Change in Muscle Sympathetic Nerve Activity (MSNA) burst incidence | Baseline, 6 weeks
  Number of bursts recorded via microneurography

SECONDARY OUTCOMES:
Change in Hot Flash Frequency | Baseline, 6 weeks
  Number of hot flashes indicated through self-reporting
Chang in sleep duration | Baseline, 6 weeks
  Measured by actigraphy data defined as recorded number of minutes in sleep
Change in wake after sleep onset | Baseline, 6 weeks
  Measured by actigraphy data defined as number of minutes from sleep onset to waking
Change in Pittsburgh Sleep Quality Index | Baseline, 6 weeks
  The Pittsburgh Sleep Quality Index measures the severity of sleep disturbances. Possible scores range from 0 to 21 with higher scores indicating a worse outcome/more severe symptoms of sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Baker, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No